CLINICAL TRIAL: NCT03170674
Title: CSD170501: A Randomized, Controlled Study to Assess Biomarkers of Tobacco Exposure in Smokers During In-Clinic Confinement Switch to an Electronic Cigarette
Brief Title: CSD170501: Study to Assess Biomarkers of Tobacco Exposure in Smokers During In-Clinic Confinement Switch to an Electronic Cigarette
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Collaborators: Vince & Associates Clinical Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSD170501
Record Dates: First submitted 2017-05-24; First posted 2017-05-31 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FT21039 Product Use Group (Experimental): Subjects will use the electronic cigarette product (FT21039).
  Interventions: Other: FT21039
- FT21092 Product Use Group (Experimental): Subjects will use the electronic cigarette product (FT21092).
  Interventions: Other: FT21092
- FT21018 Product Use Group (Experimental): Subjects will use the electronic cigarette product (FT21018).
  Interventions: Other: FT21018
- Abstinence Group (No Intervention): Subjects in the Abstinence Group will not be assigned any products.

INTERVENTIONS:
Other: FT21039 — an electronic cigarette product
  Arms: FT21039 Product Use Group
Other: FT21092 — an electronic cigarette product
  Arms: FT21092 Product Use Group
Other: FT21018 — an electronic cigarette product
  Arms: FT21018 Product Use Group

SUMMARY:
The purpose of this clinical study is to evaluate changes in biomarkers of exposure (BOE) to tobacco smoke constituents after smokers switch from combustible cigarettes to use of one of the three electronic cigarettes or abstinence.

DETAILED DESCRIPTION:
This will be a two-center, randomized, controlled, switching, open-label, parallel cohort study. The study will compare biomarkers of tobacco exposure from subjects at baseline levels of biomarkers of tobacco exposure after they have switched to one of three electronic cigarettes or abstinence for 5 days.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an Informed Consent Form (ICF) and complete questionnaires written in English;
2. Generally healthy males or females, 21 to 60 years of age (inclusive);
3. Screening expired carbon monoxide (ECO) level ≥ 12 parts per million (ppm);
4. Self-reports that cigarettes are the only tobacco or nicotine-containing product used within 30 days of the Screening Visit (Note: Rare use of other products [e.g., cigar or bridging therapy with NRT] may be acceptable in consultation with the Sponsor);
5. Self-reports at the Screening Visit smoking on average at least 10 cigarettes per day that are filtered, non-menthol, 83 mm to 100 mm length and inhaling the smoke for at least 6 months prior to the Screening Visit (Note: Smokers who use menthol cigarette products like Camel Crush are not eligible for the study);
6. Positive urine cotinine test at Screening and Enrollment;
7. Willing to switch from current cigarette to one of the Investigational Products or to abstain from smoking for approximately 7 days during in-clinic confinement;
8. Females of childbearing potential must be willing to use a form of contraception acceptable to the Investigator from the time of signing the ICF until Study Discharge or be surgically sterile for at least 90 days prior to the Screening Visit;
9. Able to safely perform the required study procedures, as determined by the Investigator.

Exclusion Criteria:

1. Clinically significant or unstable/uncontrolled acute or chronic medical conditions at screening, as determined by the Investigator, that would preclude a subject from participating safely in the study (e.g., hypertension, chronic lung disease, heart disease, neurological disease, or psychiatric disorders) based on screening assessments such as safety labs, medical history, and physical/oral examinations;
2. Self-reports or safety labs that indicate diabetes;
3. Use of medicine for treatment of depression, unless on a stable dose for the past 6 months prior to screening and deemed clinically stable by the PI.
4. Current scheduled treatment for asthma within the past consecutive 12 months prior to screening. As needed treatment, such as inhalers, may be included at the PIs discretion pending approval from the medical monitor.
5. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
6. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for 5 minutes (at Screening or Day -2 Check-in);
7. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV);
8. Clinically significant hemoglobin level, < 5% of the Lower Limit of Normal (LLN), as determined by the Investigator at Screening;
9. History or presence of hemophilia or any other bleeding or clotting disorders;
10. Use of anticoagulants (e.g., clopidogrel [Plavix®], warfarin [Coumadin®, Jantoven®], aspirin [> 325 mg/day]) at least 30 days prior to screening;
11. Given a whole blood donation within 8 weeks (≤56 days) prior to enrollment;
12. Plasma donation within ≤ 7 days prior to enrollment;
13. Weight of ≤ 110 pounds;
14. Postponing a decision to quit smoking (defined as planning a quit attempt within 30 days of Screening) to participate in this study;
15. Employed by a tobacco company, the clinical study site, or handles e-liquids or unprocessed tobacco as part of his/her job;
16. Use of any medication or supplement that aids in smoking cessation including, but not limited to, any nicotine replacement therapy (NRT) unless used for short term bridging therapy (e.g., nicotine gum, lozenge, patch), varenicline (Chantix), bupropion (Wellbutrin, Zyban), or lobelia extract within 30 days of the Screening Visit;
17. Use of injectable forms of medication(s) for the duration of the study, unless acceptable in the opinion of the Investigator or with the exception of injectable forms of birth control that are not required to be administered during the study period;
18. Self-reports drinking more than 14 servings of alcoholic beverages per week (1 serving = 12 oz of beer, 6 oz of wine, or 1.5 oz of liquor);
19. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study;
20. Females ≥35 years of age currently using systemic, estrogen-containing contraception, or hormone replacement therapy for menopause-related symptoms;
21. A positive urine drug screen without disclosure of corresponding prescribed concomitant medication(s) at the Screening Visit or Enrollment;
22. A positive alcohol test at Screening or Enrollment;
23. Regularly exposed to solvent fumes or gasoline (e.g., painter, auto mechanic);
24. Participation in another clinical study within 30 days prior to the time of consent. The 30-day window for each subject will be derived from the date of the last study event in the previous study to time of consent of the current study;
25. Determined by the Investigator to be inappropriate for this study, including a subject who is unable to communicate or unwilling to cooperate with the clinical staff;
26. Unable or unwilling to participate in the in-clinic confinement for the full study duration (total of 10 days).

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Biomarkers of Tobacco Exposure in Urine to Day 5 | 5 days
  A comparison of biomarkers of tobacco exposure in urine from subjects at baseline and for 5 days after they have switched to one of the electronic cigarette products or abstinence.
  Biomarkers of tobacco exposure in urine include:
  1. 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol) (NNAL) + glucuronides
  2. N'-nitrosonornicotine (NNN) + glucuronides
  3. 4-aminobiphenyl
  4. 1-aminonaphthalene
  5. 2-aminonaphthalene
  6. o-toluidine
  7. S-phenyl mercapturic acid (SPMA)
  8. 3-hydroxy-1-methylpropyl-mercapturic acid (HMPMA)
  9. 2-cyanoethyl mercapturic acid (CEMA)
  10. Monohydroxybutyl mercapturic acid (MHBMA)
  11. 3-hydroxypropyl mercapturic acid (HPMA)
  12. 3-hydroxy-benzo[a]pyrene
Change from Baseline Biomarkers of Tobacco Exposure in Blood to Day 5 | 5 days
  A comparison of biomarkers of tobacco exposure in blood from subjects at baseline and for 5 days after they have switched to one of the electronic cigarette products or abstinence.
  Biomarkers of tobacco exposure in blood include:
  1. Carboxyhemoglobin

SECONDARY OUTCOMES:
Change from Baseline Biomarkers of Tobacco Exposure in Urine to Day 5 | 5 days
  A comparison of biomarkers of tobacco exposure in urine from subjects at baseline and for 5 days after they have switched to one of the electronic cigarette products or abstinence.
  Biomarkers of tobacco exposure in urine include:
  1. Unconjugated nicotine
  2. Unconjugated cotinine
  3. Unconjugated trans-3'-hydroxycotinine
  4. Nicotine-N-glucuronide
  5. Cotinine-N-glucuronide
  6. Trans-3'-hydroxycotinine-O-glucuronide
Change from Baseline Biomarkers of Tobacco Exposure in Blood to Day 5 | 5 days
  A comparison of biomarkers of tobacco exposure in blood from subjects at baseline and for 5 days after they have switched to one of the electronic cigarette products or abstinence.
  Biomarkers of tobacco exposure in blood include:
  1. Plasma nicotine
  2. Plasma cotinine

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kelsh, MD, Principal Investigator — Vince & Associates Clinical Research, Inc.
Locations (2):
- United States (2):
  - Vince & Associates Clinical Research, Inc., Overland Park, Kansas
  - DaVita Clinical Research, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No